CLINICAL TRIAL: NCT07218822
Title: Impact of Pistachio Consumption on Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAAV9510
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Poor Quality Sleep
MeSH Terms: interventions — Hazard Analysis and Critical Control Points

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, dietary intervention with two intervention periods of 4 weeks each, separated by 2-4 week washout period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pistachio (Active Comparator): During the experimental (pistachio) intervention period, participants will be given 2 servings of pistachios (28 g each) to consume once in the morning (within 3 hours of wake time) and once in the evening (3-6 hours before bedtime) every day.
  Interventions: Dietary Supplement: Pistachio
- Control (Placebo Comparator): During the control food intervention period, participants will be given muffins and cookies (one serving each/day) to be consumed once in the morning (within 3 hours of wake time) and once in the evening (3-6 hours before bedtime) every day.
  Interventions: Dietary Supplement: Control food

INTERVENTIONS:
Dietary Supplement: Pistachio — 2 servings/day for 4 weeks (56 g total/day)
  Arms: Pistachio
Dietary Supplement: Control food — Muffins and cookies (no nuts), at an equivalent number of calories as the pistachio intervention, daily
  Arms: Control

SUMMARY:
Sleep is essential for life and overall health. Unfortunately, a large portion of the population in the U.S. and worldwide experience sleep deficiencies, which increase their risk for developing chronic diseases. These sleep difficulties often cause distress, leading individuals to seek various forms of treatment. Given that some drugs cause habituation and undesirable side effects, individuals often turn to over-the-counter sleep remedies. However, long-term use of over-the-counter treatments is not recommended by the American Academy of Sleep Medicine for insomnia treatment and there is currently no recommendation related to dietary management. There is a strong need to identify natural measures to improve sleep in millions of adults battling poor sleep. Diet is emerging as a potentially important modulator of sleep. Despite observational data linking greater nut intake with better sleep, and that pistachios contain a significant number of sleep-promoting compounds, no study to date has evaluated the impact of pistachio supplementation on sleep. To address this key knowledge gap, the investigators propose to conduct a randomized controlled trial to evaluate the impact of pistachio consumption, relative to a calorie-matched control food, on sleep in middle-aged adults with poor sleep and to explore underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Poor sleep quality, Pittsburgh Sleep Quality Index score >5
* BMI 20 - 29.9 kg/m^2
* Ability to abstain from travel across time zones
* Willingness to eat study foods
* Willingness/ability to discontinue use of vitamin and mineral supplements

Exclusion Criteria:

* Premenopausal women
* Medical or living conditions that could affect sleep:

  * Smoking
  * Excessive caffeine intake (>300 mg/day)
  * Non-day shift work
  * Chronic pain
  * Diagnosis of a chronic disease (e.g., uncontrolled hypertension, pre-diabetes, type 2 diabetes, chronic kidney disease, chronic obstructive pulmonary disease)
* Autoimmune diseases, cardiovascular event or cancer in the past 24 months
* Psychiatric/neurologic disease or disorder, or sleep disorder (diagnosed or high risk for sleep apnea, chronic insomnia, restless leg syndrome, narcolepsy)
* Allergy or intolerance to nuts or study foods
* Use of medications that influence CYP1A2 and selective serotonin reuptake inhibitors

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported sleep quality | 4 weeks
  Self-reported sleep quality will be reported by the score on the Pittsburgh Sleep Quality Index. The full score range is 0 to 21, where a higher score indicates worse sleep quality.
Objective sleep quality | 4 weeks
  Sleep fragmentation index assessed by wrist actigraphy. This is a measure of how frequently sleep is interrupted, calculated as the sum of the percentage of all scored epochs with one or more activity counts during time in bed and percentage of one-minute periods of sleep vs all periods of sleep during the sleep period.
Overnight melatonin production | 4 weeks
  Amount of 6-sulfatoxymelatonin present in urine collected overnight, reported as ng/mg creatinine (corrected for creatinine content).

SECONDARY OUTCOMES:
Sleep efficiency | 4 weeks
  Percent of time in bed spent asleep from wrist actigraphy
Sleep depth | 4 weeks
  Time spent in deep sleep from home sleep test
Sleepiness | 4 weeks
  Sleepiness will be reported by the score on the Epworth Sleepiness Scale. The full score range is 0 - 10, where a higher score indicates greater sleepiness.
Insomnia symptoms | 4 weeks
  Insomnia symptoms will be assessed using the Insomnia Severity Index. The full score range is 0 - 28, where a higher score indicates more severe insomnia.

OTHER OUTCOMES:
Gut microbial diversity | 4 weeks
  Shannon index of alpha-diversity
Polyphenols | 4 weeks
  Total amount of polyphenols present in urine collected overnight
Polyphenol subtypes | 4 weeks
  Amount of each polyphenol subtype detected in urine collected overnight

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided